CLINICAL TRIAL: NCT04836091
Title: A Patient-centered Decision Aid to Inform HIV Prevention Choices for At-risk Male Couples in New Relationships
Brief Title: Acceptability, Feasibility and Preliminary Impact of OurPlan, an mHealth HIV Prevention Intervention for Male Couples
Acronym: OurPlan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Dr. Jason Mitchell, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH116684 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Waiting Lists; Methods

STUDY DESIGN:
Intervention Model Description: Two-month pilot randomized controlled trial with a a waitlist control condition of one month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): From baseline to 2-month post-test, participants in the intervention arm will have access to the OurPlan program app.
  Interventions: Behavioral: Intervention
- Waitlist-delayed intervention (Experimental): Participants in this study arm will not have access to the OurPlan program in the app from baseline to day 30 (month 1) of the trial. From day 31 to day 60, participants in this study arm will be given access to the OurPlan program in the app.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Waitlist — From day 31 to day 60 (ie., during month 2) of the trial, participants in the waitlist arm will be granted access and instructed to use the OurPlan program as directed. The OurPlan program includes 4 modules covering topics of communication, HIV/STI prevention, HIV/STI statistics, and stigma / discrimination. Each module contains content, questions, and an activity for the participant and couple to complete. OurPlan also includes a resource locator using GPS-capabilities to allow participants to find sexual health resources, as well as a calendar and reminder system. One goal of OurPlan is to help both partners of the couple create and use a risk-reduction plan of evidence-based prevention strategies over time. Answers provided during the assessments will help determine whether participants/couples created a risk-reduction plan and used evidence-based strategies over time, including changes in their own and partner-related attitudes toward these strategies.
  Arms: Waitlist-delayed intervention
Behavioral: Intervention — From day 1 to day 60 (ie., entire 2 month duration) of the trial, participants in the intervention arm will be granted access and instructed to use the OurPlan program as directed. The OurPlan program includes 4 modules covering topics of communication, HIV/STI prevention, HIV/STI statistics, and stigma / discrimination. Each module contains content, questions, and an activity for the participant and couple to complete. OurPlan also includes a resource locator using GPS-capabilities to allow participants to find sexual health resources, as well as a calendar and reminder system. One goal of OurPlan is to help both partners of the couple create and use a risk-reduction plan of evidence-based prevention strategies over time. Answers provided during the assessments will help determine whether participants/couples created a risk-reduction plan and used evidence-based strategies over time, including changes in their own and partner-related attitudes toward these strategies.
  Arms: Immediate intervention

SUMMARY:
The study will evaluate the use and preliminary impact of an mHealth app for improving sexual health outcome measures among male couples by assessing whether exposure and use of the app results in improvements in participants and couples' self-reported sexual health and prevention behaviors, beliefs, and attitudes. The study will enroll both men of the couple into a randomized controlled trial. Participants/couples randomized to the intervention will have access to the app for two months while those assigned to the waitlist group will receive and have access to the app for one month. Participants will complete surveys at baseline and at month 2.

DETAILED DESCRIPTION:
The study will evaluate the use and preliminary impact of an mHealth app for improving sexual health outcome measures among male couples by assessing whether exposure and use of the app results in improvements in participants and couples' self-reported sexual health and prevention behaviors, beliefs, and attitudes. The study will enroll both partners of the 42 male couples into a 2-month randomized controlled trial with a waitlist control condition of one month. Couples will be assigned to either the immediate intervention group ("intervention arm") or the waitlist-control group ("waitlist-control arm"). All participants will take an assessment survey at baseline, and the intervention group will be oriented on the installation and use of the app upon randomization to that group. The waitlist-control group will follow the same procedures one month later. Participants/couples randomized to the intervention arm will have access to the intervention app for two months (ie, day 1-60) while those assigned to the waitlist-control group will have access to the app for one month (ie, day 31-60). All participants in the randomized controlled trial will complete a short follow-up survey at month 2 and a brief exit interview.

ELIGIBILITY:
Inclusion Criteria for both partners of the male couple:

* self-reported that currently self-identifies as a male
* self-reported in a sexual relationship with another self-identified male
* self-reported relationship length between 1 and 12 months
* self-reported anal sex with relationship partner in past 2 months
* owns and uses an Internet-connected smartphone or tablet
* resides in the U.S.
* self-reported ability to read and understand English-language

Exclusion Criteria:

* Does not meet one or more the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans men and cisgender men
Enrollment: 84 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in presence of a detailed risk-reduction plan | Baseline, month 2
  Men will be asked if they created a detailed risk-reduction plan containing evidence-based strategies of routine HIV/STI testing, consistent condom use, PrEP, and ART
Change in number of evidence-based prevention strategies being used over time | Baseline, month 2
  Men will be asked how many evidence-based HIV/STI prevention strategies they are currently using
Change in willingness to use evidence-based prevention strategies over time | Baseline, month 2
  Men will be asked about their willingness to use evidence-based prevention strategies
Change in intention to use evidence-based prevention strategies over time | Baseline, month 2
  Men will be asked about their intention to use evidence-based prevention strategies

SECONDARY OUTCOMES:
Change in HIV transmission and prevention knowledge | Baseline, month 2
  Men will be asked about their knowledge on HIV transmission and prevention over time
Change in goal congruence on sexual health | Baseline, month 2
  Men will be asked about their goal congruence regarding sexual health and their relationship partner
Change in mutual constructive communication | Baseline, month 2
  Men will be asked about their mutual constructive communication patterns over time

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Interested researchers must email the PI with a request to access de-identified, anonymous IPD. The PI will review such requests for secondary analyses using de-identified data that have already been published.